CLINICAL TRIAL: NCT03759925
Title: Food as Medicine: Providing Medically Appropriate Meals to Patients After Discharge for Congestive Heart Failure Exacerbation
Brief Title: Cardiac Recovery Through Dietary Support
Acronym: CaRDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); San Francisco General Hospital (Other); Project Open Hand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-20742
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Nutritional Support

STUDY DESIGN:
Intervention Model Description: 180 participants will be randomized to the intervention (n=90) or control (n=90) groups, stratified by health care utilization (<3 vs. >=3 hospital admissions at ZSFGH) and food security ( zero affirmative answers vs. at least one affirmative answers on the US Department of Agriculture (USDA) 12-question food security screener). The intervention consists of providing home delivery of medically-appropriate food support and individual nutritional counseling over five months to patients at Zuckerberg San Francisco General admitted to the hospital with acute decompensated heart failure.
Who Masked: Investigator
Masking Description: The principal investigators will be masked to whether participants were in the intervention or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Support (Experimental): The intervention consists of home delivery of medically-appropriate food support (DASH and diabetic diet compliant) in the form of prepared meals and/or groceries and monthly individual nutritional counseling with a Registered Dietician.
  Interventions: Other: Nutritional Support
- Standard of Care (No Intervention): The control group will receive standard of care follow up care after their hospitalization for acute decompensated heart failure.

INTERVENTIONS:
Other: Nutritional Support — Weekly nutritional components: Month 1: equivalent of 3 meals/day in the form of 14 frozen meals, and breakfast bag with items to prepare 7 breakfast meals. Month 2: equivalent of 3 meals a day in the form of 7 frozen meals, grocery bags, and breakfast bags with items to prepare 7 breakfast meals. Month 3: the equivalent of 2 meals a day in the form of 7 frozen meals and grocery bags. Month 4: Participant choice to receive either 7 frozen meals or grocery bag with equivalent food for 1 meal a day. Month 5: Grocery bag with equivalent food for 1 meal a day Nutritional counseling component: Individual counseling with Registered Dietician monthly
  Arms: Nutritional Support

SUMMARY:
This is a prospective, randomized, wait-list controlled study examining the impact of providing medically appropriate meals to patients discharged from Zuckerberg San Francisco General Hospital after acute decompensated heart failure. Upon discharge, patients will be randomized to either the intervention or wait list control arm. The intervention is the delivery of medically appropriate meals and groceries to patients' homes in a tapered manner over five months (the equivalent of three meals a day for 60 days, then the equivalent of two meals a day for 30 days, then the equivalent of one meal a day for 60 days) and monthly assessments with a registered dietician (RD). All food and RD assessments are administered via a community partner, Project Open Hand, as a modification of current offerings for clients at Project Open Hand. Subjects randomized into the wait list control arm will receive the food intervention five months after discharge. The study's primary aim is to examine the impact of nutritional support on the Kansas City Cardiomyopathy Questionnaire scores. In addition, the study aims to examine the impact of nutritional support on healthcare utilization (particularly readmission rates and emergency room utilization), dietary change, medication adherence, and quality of life.

DETAILED DESCRIPTION:
The San Francisco Department of Public Health, University of California at San Francisco (UCSF), and Project Open Hand (POH), a community based organization in San Francisco which provides meals and groceries to chronically ill clients in the Bay Area, have partnered to conduct a prospective, randomized, wait-list controlled study examining the impact of providing medically appropriate meals and registered dietician (RD) support to patients discharged from Zuckerberg San Francisco General Hospital after acute decompensated heart failure. Before discharge, patients will be randomized to either the intervention or wait list control arm. The intervention consists of the delivery of medically appropriate meals and/or groceries to participants' homes in a tapered manner over five months (the equivalent of three meals a day for 60 days, then the equivalent of two meals a day for 30 days, then the equivalent of one meal a day for 60 days) and monthly nutrition education with a registered dietician (RD). All food and nutritional education are administered by POH staff and RDs. Participants randomized into the wait list control arm will receive the food intervention five months after discharge. The study's primary aim is to examine the impact of nutritional support on the Kansas City Cardiomyopathy Questionnaire scores. In addition, the study aims to examine the impact of nutritional support on healthcare utilization (particularly readmission rates and emergency room utilization), dietary change, medication adherence, and quality of life. The investigators will assess outcomes at baseline while patients are hospitalized, 1 month after discharge, and 5 months after discharge using quantitative surveys. The investigators will call participants at 3 months and 4 months after discharge with a shorter quantitative survey assessing a subset of outcome measures. In addition, the investigators will conduct a qualitative interview near the conclusion of the intervention in a subset of participants to understand perceived impacts of the intervention as well as barriers and facilitators to heart failure care.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized at Zuckerberg San Francisco General Hospital (ZSFG) with acute decompensated heart failure/congestive heart failure exacerbation
* Adults with their primary residence within San Francisco
* Age: >18 years old
* Languages: English or Spanish
* Housed at a location where they would be able to securely receive, store and reheat food

Exclusion Criteria:

* Patients with severe or critical aortic stenosis.
* Patients with six or more hospital admissions within the last twelve months
* Patients who are being discharged to a living facility that provides meals to residents.
* Patients who anticipate moving from their current housing situation to one that does not meet our inclusion criteria within six months of enrollment.
* Patients who are part of meal provision program that provides more than 7 meals a week to the patient.
* Patients who are unable to feed themselves and do not have adequate support to help them with feeding.
* Patients with limited physical, cognitive, or behavioral abilities that would interfere with their ability to follow-up with a study as determined by their ability to receive the Project Open Hand services and follow up with survey interviews
* Patients with anticipated life expectancy of less than a year.
* Patients who lack capacity to consent to a research study.
* Patients currently requiring dialysis or determined to be in need of dialysis in the next 6 months.
* Patients with severe allergies to eggs, soy, wheat, nuts, seeds, seed oils, pineapple, raisins, or certain vegetables such as onions (allergies are considered on a case-by-case basis in consultation with Project Open Hand).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Change in the overall Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to one month by study arm | Baseline and one month
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.The change in the overall score from baseline to one month will be reported.
Change in the overall Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to five months by study arm | Baseline and five months
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. The change in the overall score from baseline to five months will be reported.
Change in the clinical summary Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to one month by study arm | Baseline and one month
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. A clinical summary score can be obtained from the symptom frequency and burden domains and the physical limitation domain. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.The change in the clinical summary score from baseline to one month will be reported by study arm.
Change in the clinical summary Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to five months by study arm | Baseline and five months
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. A clinical summary score can be obtained from the symptom frequency and burden domains and the physical limitation domain. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.The change in the clinical summary score from baseline to five months will be reported by study arm.
Change in the physical domain Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to one month by study arm | Baseline and one month
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores from the physical domain can be transformed to 0 to 100 , in which higher scores reflects better health status.The change in the physical domain score from baseline to one month will be reported by study arm.
Change in the physical domain Kansas City Cardiomyopathy Questionnaire (KCCQ) scores from baseline to five months by study arm | Baseline and five months
  The Kansas City Cardiomyopathy Questionnaire is a 23-item instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores from the physical domain can be transformed to 0 to 100 , in which higher scores reflects better health status.The change in the physical domain score from baseline to five months will be reported by study arm.

SECONDARY OUTCOMES:
Hospital admissions from baseline to 1 month, by study arm | Baseline and 1 month
  Number of admissions to hospitals that is a composite of: 1) At baseline, participants will self-report ER visits to hospitals OTHER than Zuckerberg San Francisco General Hospital in the past three months, and 2) the number of admissions to Zuckerberg San Francisco General will be determined by medical records. The number of hospital admissions from baseline to 1 month after discharge, by study arm will be reported.
Hospital admissions from baseline to 5 month, by study arm | Baseline and 5 months
  Number of admissions to hospitals that is a composite of:1) At baseline, participants will self-report ER visits to hospitals OTHER than Zuckerberg San Francisco General Hospital in the past three months, and 2) the number of admissions to Zuckerberg San Francisco General will be determined by medical records. The number of hospital admissions from baseline to five month after discharge, by study arm will be reported.
Emergency room utilization at any hospital from baseline to 1 month, by study arm. | Baseline and 1 month
  Number of emergency room visits that is a composite of: 1) At baseline, participants will self-report emergency room visits to hospitals OTHER than Zuckerberg San Francisco General Hospital in the past three months, and 2) the number of emergency room visits at Zuckerberg San Francisco General will be determined by medical records.The number of emergency room visits will be reported from baseline to 1 month after discharge, by study arm.
Emergency room utilization at any hospital from baseline to 5 month, by study arm. | Baseline and 5 months
  Number of ER visits that is a composite of: 1) At baseline, participants will self-report emergency room visits to hospitals OTHER than Zuckerberg San Francisco General Hospital in the past three months, and 2) the number of emergency room visits at Zuckerberg San Francisco General will be determined by medical records.The number of emergency room visits admissions will be reported from baseline to 1 month after discharge, by study arm.
Change in overall health-related quality of life from baseline to five months, by study arm | Baseline and five months
  Health-related quality of life will be measured using the 4-item Healthy Days Core Module of the Center for Disease Control and Prevention's (CDC) Health-Related Quality of Life survey. This module asks the number of days in the past 30 days the person felt physically or mentally unwell. The summary index then estimates the number of healthy days subtracting the number of unhealthy days from 30 days. The change in healthy days from baseline to five months by study arm will be reported.
Change in food insecurity severity from baseline to one month by study arm | Baseline and 1 month
  The 10-item adult version of the US household food security survey module from the US Department of Agriculture (USDA) will be used to assess the change in the food security scores from baseline to one month. The score ranges from 0 to 18 in households with children, and 0 to 10 in households without children. Higher score indicates higher severity of food insecurity. The change in the food insecurity scores from baseline to one month by study arm will be reported.
Change in food insecurity severity from baseline to five months by study arm | Baseline and 5 months
  The 10-item adult version of the US household food security survey module from the US Department of Agriculture (USDA) will be used to assess the change in the food security scores from baseline to five months. The score ranges from 0 to 18 in households with children, and 0 to 10 in households without children. Higher score indicates higher severity of food insecurity. The change in the food insecurity scores from baseline to five months by study arm will be reported.
Change in consumption of food high in sodium from baseline to five months by study arm. | Baseline and five moths
  Food consumption was collected using food frequency questionnaire that assess the frequency of intake of 32 food items in the prior month. A change in the consumption (servings/day) of food high in sodium from baseline to five months will be reported.
Change in consumption of food high in saturated fat consumption from baseline to five months by study arm. | Baseline and five months
  Food consumption was collected using food frequency questionnaire that assess the frequency of intake of 32 food items in the prior month. A change in the consumption (servings/day) of food high in saturated fat from baseline to five months will be reported.
Change in medication adherence from baseline to five months, by study arm | Baseline and five months
  A Single-Item Rating Visual Analogue Scale (range 0-100) for medication adherence will estimate the percentage of medications taken in the past month and is reliable and valid, including in low-literacy populations. A higher value indicates higher adherence. The change in medication adherence (percentage points) from baseline to five months between intervention and control arms will be reported.
Change in depressive symptoms from baseline to five months, by study arm | Baseline and five months
  Change in depressive symptoms, using the 9 items Patient Health Questionnaire (PHQ-9), with scores ranging from 0 to 27, with higher scores indicating higher levels of depression. The change in PHQ-9 scores from baseline to one month, and from baseline to five months among by study arms will be reported.

OTHER OUTCOMES:
Hospital admissions to Zuckerberg San Francisco General Hospital from baseline to nine months, by study arm | Baseline and nine months
  Number of admissions to Zuckerberg San Francisco General Hospital as determined by the medical records from baseline to one month, by study arm will be reported.
Emergency room utilization utilization at Zuckerberg San Francisco General Hospital from baseline to nine months by study arm | Baseline and nine months
  Number of Emergency Room visits at Zuckerberg San Francisco General Hospital as determined by the medical records will be reported by study arm from baseline to nine months.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nguyen, MD, Principal Investigator — San Francisco Department of Public Health, UCSF; Sheri Weiser, MD, MPH, MA, Principal Investigator — University of California, San Francisco; Kartika Palar, PhD, Principal Investigator — University of California, San Francisco; Binh An Phan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell AD, Godfryd A, Buys DR, Locher JL. Does Participation in Home-Delivered Meals Programs Improve Outcomes for Older Adults? Results of a Systematic Review. J Nutr Gerontol Geriatr. 2015;34(2):124-67. doi: 10.1080/21551197.2015.1038463. PMID 26106985
- [Background] Ford ES. Food security and cardiovascular disease risk among adults in the United States: findings from the National Health and Nutrition Examination Survey, 2003-2008. Prev Chronic Dis. 2013 Dec 5;10:E202. doi: 10.5888/pcd10.130244. PMID 24309090
- [Background] Gurvey J, Rand K, Daugherty S, Dinger C, Schmeling J, Laverty N. Examining health care costs among MANNA clients and a comparison group. J Prim Care Community Health. 2013 Oct;4(4):311-7. doi: 10.1177/2150131913490737. Epub 2013 Jun 3. PMID 23799677
- [Background] Seligman HK, Jacobs EA, Lopez A, Tschann J, Fernandez A. Food insecurity and glycemic control among low-income patients with type 2 diabetes. Diabetes Care. 2012 Feb;35(2):233-8. doi: 10.2337/dc11-1627. Epub 2011 Dec 30. PMID 22210570
- [Background] Seligman HK, Lyles C, Marshall MB, Prendergast K, Smith MC, Headings A, Bradshaw G, Rosenmoss S, Waxman E. A Pilot Food Bank Intervention Featuring Diabetes-Appropriate Food Improved Glycemic Control Among Clients In Three States. Health Aff (Millwood). 2015 Nov;34(11):1956-63. doi: 10.1377/hlthaff.2015.0641. PMID 26526255
- [Background] Weiser SD, Hatcher A, Frongillo EA, Guzman D, Riley ED, Bangsberg DR, Kushel MB. Food insecurity is associated with greater acute care utilization among HIV-infected homeless and marginally housed individuals in San Francisco. J Gen Intern Med. 2013 Jan;28(1):91-8. doi: 10.1007/s11606-012-2176-4. Epub 2012 Aug 18. PMID 22903407
- [Background] Zilak, J.P. & Gunderson, C. (2014). The health consequences of senior hunger in the United States: Evidence from the 1999-2010 NHANES. Retrieved from: http://www.humsenior.org/dmdocuments/Senior%20Hunger_article.pdf?lbisphpreq=1

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03759925/Prot_SAP_000.pdf